CLINICAL TRIAL: NCT05018728
Title: The Effect of Voxelotor on Cerebral Hemodynamic Response in Children With Sickle Cell Anemia
Acronym: VoxSCAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated on September 26, 2024 due to voluntary withdrawal of study drug from the market.
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002483
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Anemia in Children
MeSH Terms: interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voxelotor (Experimental): Children with sickle cell anemia taking voxelotor for 12 weeks.
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — Voxelotor is taken orally once a day. Participants 12 years or older will take 1500 mg/day. Participants younger than 12 years of age will receive a dose based on their body weight to provide exposure corresponding to the adult dose of 1500 mg/day.
  Other Names: Oxbryta

SUMMARY:
Voxelotor is a new drug for adolescents and adults with sickle cell disease that improves hemoglobin levels and reduces the incidence of worsening anemia. However, it is unclear whether this increase in hemoglobin is associated with a reduction in cerebral metabolic stress. This study will measure the effects of voxelotor on cerebral hemodynamics.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a genetic blood disorder that has profound effects on the brain. In the presence of chronic anemia, the brain microvasculature dilates in order to maintain adequate oxygen delivery to the tissue. As cerebral blood flow increases and the vasculature becomes maximally dilated, oxygen extraction fraction (OEF) increases to keep up with metabolic demand. Unfortunately, this state of maximized response leaves the brain vulnerable and ill-equipped to adapt to increased metabolic demand; consequently, the tissue is susceptible to infarction when blood flow/volume are insufficient to maintain sufficient oxygen metabolism.

Voxelotor is a first-in-class drug approved by the FDA for treatment of adults and children (aged four years and older) with SCD. This study will examine the effects of voxelotor on cerebral hemodynamics. The researchers hypothesize that as hemoglobin increases due to voxelotor, cerebral blood flow and oxygen extraction fraction will decrease. To test this hypothesis, measurements of brain blood flow, oxygen extraction, and oxygen metabolism will be made using a customized diffuse correlation spectroscopy and frequency domain near-infrared spectroscopy system (DCS/fdNIRS). This non-invasive, optical technique uses light to estimate an average oxygen saturation of the microvasculature, i.e., capillaries, arterioles, and venules.

All participants will receive voxelotor, administered orally once daily as tablets, dispersible tablets or as powder for oral suspension at a dose based on their body weight, for 12 weeks. Measurements of cerebral blood flow, oxygen extraction, and oxygen metabolism will be made at baseline (before starting drug), and at 4, and 12 weeks after the start of voxelotor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed parental/guardian consent and participant assent/consent has been obtained per institutional review board (IRB)/Ethics Committee (EC) policy and requirements, consistent with International Conference on Harmonization (ICH) guidelines
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female participants, ages 4 to 30 years, inclusive
* Homozygous hemoglobin SS (HbSS) or hemoglobin S/beta^0 thalassemia (HbS/β^0 thal)
* Hemoglobin (Hb) ≤10.5 g/dL at baseline
* Concomitant hydroxyurea (HU) therapy is allowed if the dose has been stable for at least 3 months with no anticipated need for dose adjustments during the study and no sign of hematological toxicity
* Ability to take oral medication and willingness to adhere to daily voxelotor and scheduled DCS/NIRS assessments
* If sexually active and female, must agree to abstain from sexual intercourse or to use a highly effective method of contraception throughout the study period and for 30 days after discontinuation of study drug. If sexually active and male, must agree to abstain from sexual intercourse or willing to use barrier methods of contraception throughout the study period and for 30 days after discontinuation of study drug.
* Females of child-bearing potential, i.e., who have begun menstruation and are sexually active, are required to have a negative pregnancy test at screening before the initial administration of study drug.

Exclusion Criteria:

* Any one of the following requiring medical attention within 14 days prior to signing the informed consent form (ICF):

  * Vaso-occlusive crisis (VOC)
  * Acute chest syndrome (ACS)
  * Splenic sequestration crisis
  * Dactylitis
* Requires chronic transfusion therapy
* Red blood cell (RBC) transfusion within 60 days of signing the ICF
* Renal dysfunction requiring chronic dialysis or creatinine ≥1.5 mg/dL
* Hepatic dysfunction characterized by alanine aminotransferase (ALT) >4× upper limit of normal (ULN) for age
* Clinically relevant cardiac abnormality, in the opinion of the Investigator, such as:

  * Hemodynamically significant heart disease, e.g., congenital heart defect, uncompensated heart failure, or any unstable cardiac condition
  * An arrhythmic heart condition requiring medical therapy
* Corrected QT interval by Fridericia (QTcF) >450 msec, congenital long QT syndrome, second- or third-degree heart block at rest (with the exception of asymptomatic Mobitz type I second degree heart block)
* Received an investigational drug within 30 days or 5 half-lives, whichever is longer, of signing the ICF
* Heavy smoker (defined as smoking more than 10 cigarettes/day or its nicotine equivalent including e-cigarettes)
* Unlikely to comply with the study procedures
* Other medical, psychological, or addictive condition that, in the opinion of the Investigator, would confound or interfere with evaluation of safety and/or pharmacokinetics (PK) of the investigational drug, prevent compliance with the study protocol, or preclude informed consent
* Any condition affecting drug absorption, such as major surgery involving the stomach or small intestine (prior cholecystectomy is acceptable)
* History of malignancy within the past 2 years prior to treatment Day 1 requiring chemotherapy and/or radiation (with the exception of local therapy for non-melanoma skin malignancy)
* Clinically significant bacterial, fungal, parasitic, or viral infection currently receiving or that will require therapy

  * Participants with acute bacterial infection requiring antibiotic use should delay screening until the course of antibiotic therapy has been completed and the infection has resolved, in the opinion of the investigator
  * Known active hepatitis A, B, or C infection or human immunodeficiency virus (HIV)-positive; known active
  * Known active malaria
* Pregnant patients
* Evidence of abnormal high blood flow velocities on transcranial doppler (TCD) of 200 cm/sec or more

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow (CBF) | Baseline, Weeks 4 and 12
  CBF will be measured by diffuse correlation spectroscopy and frequency domain near-infrared spectroscopy (DCS/FDNIRS).
Change in oxygen extraction fraction (OEF) | Baseline, Weeks 4 and 12
  OEF will be measured by DCS/FDNIRS. OEF is defined as the difference between arterial and venous oxygen content and it increases to keep up with metabolic demand.
Change in cerebral metabolic rate of oxygen (CMRO2) | Baseline, Weeks 4 and 12
  CMRO2 will be measured by DCS/FDNIRS. CMRO2 is the rate that the brain consumes oxygen and is a marker of brain health.

SECONDARY OUTCOMES:
Change in total hemoglobin | Baseline, Weeks 4 and 12
  Total hemoglobin levels will be assessed and the correlation between changes in CBF, OEF and CMRO2 and change in hemoglobin at 4 and 12 weeks will be evaluated.
Change in RBC content of voxelotor-modified hemoglobin | Baseline, Weeks 4 and 12
  RBC levels in voxelotor-modified hemoglobin will be assessed and the correlation between changes in CBF, OEF and CMRO2 and change in voxelotor-modified hemoglobin at 4 and 12 weeks will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tang, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Aflac Sickle Cell Comprehensive Clinics at Children's Healthcare of Atlanta, Scottish Rite, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publication of this study (text, tables, figures, and appendices) will be made available for sharing, after de-identification
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing immediately following publication, with no end date.
Access Criteria: Data will be made available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the approved proposal. Proposals should be directed to erin.buckley@emory.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Brothers RO, Turrentine KB, Akbar M, Triplett S, Zhao H, Urner TM, Goldman-Yassen A, Jones RA, Knight-Scott J, Milla SS, Bai S, Tang A, Brown RC, Buckley EM. The influence of voxelotor on cerebral blood flow and oxygen extraction in pediatric sickle cell disease. Blood. 2024 May 23;143(21):2145-2151. doi: 10.1182/blood.2023022011. PMID 38364110

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT05018728/Prot_SAP_000.pdf